CLINICAL TRIAL: NCT06806644
Title: The Role of Ultrasonography in Predicting Outcomes of Fetal Nephropathy
Acronym: FUS-IRC
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: FUS-IRC
Record Dates: First submitted 2024-12-30; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-10

CONDITIONS: Nephropathy
Keywords: Fetal nephropathy
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Congenital anomalies of the kidneys and urinary tract are among the most frequently ultrasound-indentified malformations in the prenatal period.

Thanks to the introduction of fetal ultrasound in pregnancy screening programs, the diagnosis of these abnormalities in utero allows early manegement. In fact, prenatal diagnosis allows evolutionary control of the pathology and appropriate counseling, putting in place the best therapeutic strategies at birth. However, the predictive value of prenatal ultrasound findings is often difficult to establish.

Therefore, the investigators want to evaluate the postnatal outcomes in fetuses prenatally diagnosed with unilateral nephropathy, specifically the rate of live births, gestational age at delivery, neonatal weight, and the need for admission of the infant to the neonatal intensive care unit (NICU).

The data collected will allow investigators to assess postnatal outcomes in fetuses prenatally diagnosed with unilateral nephropathy, identifying the prenatal ultrasound findings most associated with poor postnatal prognosis to define the role of ultrasonography in predicting outcomes of fetal nephropathy.

DETAILED DESCRIPTION:
Clinical data of single-pregnancy patients who were referred to the Pregnancy at Risk Outpatient Clinics of our center between 2007 and 2023 will be considered.

These patients were evaluated with serial ultrasound checks at the outpatient clinics for the presence of suspected unilateral nephropathy that emerged during morphologic ultrasound performed between the 19th and 21st weeks of gestation. Therefore, we will analyze the ultrasound data that emerged during serious outpatient checkups, the delivery data of patients who delivered at our center, and the postnatal data of newborns.

Information on the following will be collected for each patient:

* Age
* Type of suspected nephropathy (pyelectasis, hydronephrosis/hydroureteronephrosis, multicystic kidney, dysplasia)
* Gestational age at the time of suspected diagnosis
* Gestational age at the time of diagnosis
* Assessment of amniotic fluid
* Centile of affected kidney (<5°, normal, >95°)
* Centile of unaffected kidney (<5°, normal, >95°)
* Presence of associated abnormalities in the other anatomical districts
* Performance of invasive prenatal diagnostic methods (Karyotype analysis and CGH-array)
* Progression of nephropathy
* Involvement of contralateral kidney
* Gestational age at the time of delivery
* Mode of delivery (vaginal/caesarean section)
* Sex of the newborn at birth
* Infant's weight at birth
* Ph of newborn at birth
* APGAR index at 5 and 10 minutes
* Possible admission to neonatal intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy
* Age greater than or equal to 18 years
* Detection of Unilateral Renal Abnormalities during Confidential Ultrasound
* Delivery performed at the O.U. of Obstetrics and Prenatal Age Medicine
* Acquisition of informed consent form

Exclusion Criteria:

* Request for voluntary termination of pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients evaluated with serial ultrasound checks at the outpatient clinics of this center for the presence of risk factors for unilateral fetal nephropathy will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of rate of live births, gestational age at delivery, neonatal weight, and need for admission of the newborn to the neonatal intensive care unit (NICU). | After delivery
  For quantitative continuous type variables, the intraclass correlation coefficient (ICC) will be used, and for dichotomous variables, Cohen's k test will be used.
  For the variables considered in the study, parametric or nonparametric tests will be used according to their distribution. Quantitative variables will be analyzed with Student's t-test and/or Mann-Whitney test for comparison between the two groups. Qualitative variables, on the other hand, will be analyzed by comparison of proportions and KaplanMeier algorithm with related Log Rank test.
  Cox regression will be used to assess the possible effect of covariates and confounding factors on the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluigi Pilu, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy